CLINICAL TRIAL: NCT00797290
Title: A Clinical Outcomes Protocol of Photon/Proton Beam Radiation Therapy for Carcinoma of the Nasopharynx
Brief Title: Photon/Proton Radiation Therapy for Carcinoma of the Nasopharynx
Acronym: NP01
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment, Feasibility issues
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: UFPTI 0605-NP01
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Nasopharynx Cancer
Keywords: Nasopharynx Cancer, Proton Radiation, Outcomes
MeSH Terms: conditions — Nasopharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Photon/Proton Radiation Therapy: Photon/Proton Radiation Therapy

SUMMARY:
The purpose of this study is to collect outcomes information to see what effects photon/proton beam radiation has on nasopharynx cancer.

DETAILED DESCRIPTION:
Data collection will be obtained from the patient's medical records including initial evaluation, pathology report, dosimetry information, radiotherapy completion records and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Nasopharynx cancer.

Exclusion Criteria:

* Evidence of distant metastasis.
* Previous radiation for head and neck cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at radiaton oncology clinic
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2008-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Collect and analyze morbidity outcomes | After radiation therapy, every 4 months for at least 10 years

SECONDARY OUTCOMES:
Collect and analyze tumor control outcomes | 12 months and 24 months after radiation therapy then annually for 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Roi Dagan, MD, MS, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanguineti G, Geara FB, Garden AS, Tucker SL, Ang KK, Morrison WH, Peters LJ. Carcinoma of the nasopharynx treated by radiotherapy alone: determinants of local and regional control. Int J Radiat Oncol Biol Phys. 1997 Mar 15;37(5):985-96. doi: 10.1016/s0360-3016(97)00104-1. PMID 9169804
- [Background] Bailet JW, Mark RJ, Abemayor E, Lee SP, Tran LM, Juillard G, Ward PH. Nasopharyngeal carcinoma: treatment results with primary radiation therapy. Laryngoscope. 1992 Sep;102(9):965-72. doi: 10.1288/00005537-199209000-00002. PMID 1518360
- [Background] Fandi A, Altun M, Azli N, Armand JP, Cvitkovic E. Nasopharyngeal cancer: epidemiology, staging, and treatment. Semin Oncol. 1994 Jun;21(3):382-97. No abstract available. PMID 8209270
- [Background] Teo PM, Chan AT, Lee WY, Leung TW, Johnson PJ. Enhancement of local control in locally advanced node-positive nasopharyngeal carcinoma by adjunctive chemotherapy. Int J Radiat Oncol Biol Phys. 1999 Jan 15;43(2):261-71. doi: 10.1016/s0360-3016(98)00383-6. PMID 10030248
- [Background] Al-Sarraf M, LeBlanc M, Giri PG, Fu KK, Cooper J, Vuong T, Forastiere AA, Adams G, Sakr WA, Schuller DE, Ensley JF. Chemoradiotherapy versus radiotherapy in patients with advanced nasopharyngeal cancer: phase III randomized Intergroup study 0099. J Clin Oncol. 1998 Apr;16(4):1310-7. doi: 10.1200/JCO.1998.16.4.1310. PMID 9552031
- [Background] Cooper JS, Lee H, Torrey M, Hochster H. Improved outcome secondary to concurrent chemoradiotherapy for advanced carcinoma of the nasopharynx: preliminary corroboration of the intergroup experience. Int J Radiat Oncol Biol Phys. 2000 Jul 1;47(4):861-6. doi: 10.1016/s0360-3016(00)00558-7. PMID 10863053
- [Background] Mendenhall WM, Riggs CE Jr, Cassisi NJ: Treatment of head and neck cancers. In: DeVita VT Jr, Hellman S, Rosenberg SA, eds.: Cancer: Principles and Practice of Oncology. 7th ed. Philadelphia, Pa: Lippincott Williams & Wilkins, 2005., pp 662-732.
- [Background] Laramore GE, ed.: Radiation Therapy of Head and Neck Cancer. Berlin: Springer-Verlag, 1989.
- [Background] Cummings CW, Fredrickson JM, Harker LA, et al.: Otolaryngology - Head and Neck Surgery. Saint Louis, Mo: Mosby-Year Book, Inc., 1998.
- [Background] Marks JE, Bedwinek JM, Lee F, Purdy JA, Perez CA. Dose-response analysis for nasopharyngeal carcinoma: an historical perspective. Cancer. 1982 Sep 15;50(6):1042-50. doi: 10.1002/1097-0142(19820915)50:63.0.co;2-y. PMID 7104948
- [Background] Vikram B, Mishra UB, Strong EW, Manolatos S. Patterns of failure in carcinoma of the nasopharynx: I. Failure at the primary site. Int J Radiat Oncol Biol Phys. 1985 Aug;11(8):1455-9. doi: 10.1016/0360-3016(85)90332-3. PMID 3926733
- [Background] Xia P, Fu KK, Wong GW, Akazawa C, Verhey LJ. Comparison of treatment plans involving intensity-modulated radiotherapy for nasopharyngeal carcinoma. Int J Radiat Oncol Biol Phys. 2000 Sep 1;48(2):329-37. doi: 10.1016/s0360-3016(00)00585-x. PMID 10974445
- [Background] Lee N, Xia P, Quivey JM, Sultanem K, Poon I, Akazawa C, Akazawa P, Weinberg V, Fu KK. Intensity-modulated radiotherapy in the treatment of nasopharyngeal carcinoma: an update of the UCSF experience. Int J Radiat Oncol Biol Phys. 2002 May 1;53(1):12-22. doi: 10.1016/s0360-3016(02)02724-4. PMID 12007936
- [Background] Parsons JT, Bova FJ, Fitzgerald CR, Mendenhall WM, Million RR. Radiation optic neuropathy after megavoltage external-beam irradiation: analysis of time-dose factors. Int J Radiat Oncol Biol Phys. 1994 Nov 15;30(4):755-63. doi: 10.1016/0360-3016(94)90346-8. PMID 7960976
- [Background] Parsons JT, Bova FJ, Fitzgerald CR, Mendenhall WM, Million RR. Radiation retinopathy after external-beam irradiation: analysis of time-dose factors. Int J Radiat Oncol Biol Phys. 1994 Nov 15;30(4):765-73. doi: 10.1016/0360-3016(94)90347-6. PMID 7960977
- [Background] Bhandare N, Monroe AT, Morris CG, Bhatti MT, Mendenhall WM. Does altered fractionation influence the risk of radiation-induced optic neuropathy? Int J Radiat Oncol Biol Phys. 2005 Jul 15;62(4):1070-7. doi: 10.1016/j.ijrobp.2004.12.009. PMID 15990010